CLINICAL TRIAL: NCT03798691
Title: A Pilot Study Evaluating Immunogenicity of Herpes Zoster Subunit Vaccine in Inflammatory Bowel Disease Patients Treated With Vedolizumab
Brief Title: Immunogenicity of Herpes Zoster Subunit Vaccine in Inflammatory Bowel Disease Patients Treated With Vedolizumab
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2018-1037; SMPH/MEDICINE/GASTROENT (Other: UW Madison); A534250 (Other: UW Madison); Protocol Version 11/16/2022 (Other: UW Madison)
Record Dates: First submitted 2019-01-02; First posted 2019-01-10 (Actual); Results first posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis; Herpes Zoster
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative; Herpes Zoster

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anti-TNF monotherapy (Active Comparator): Patients with IBD on Anti-TNF monotherapy will be given the shingrix vaccine. Dose and Schedule: Two doses (0.5 mL each) administered intramuscularly according to the following schedule: A first dose at Month 0 followed by a second dose administered anytime between 2 and 6 months later.
  Interventions: Biological: Shingrix
- Vedolizumab (Active Comparator): Patients with IBD on vedolizumab monotherapy will be given the shingrix vaccine.
  Dose and Schedule: Two doses (0.5 mL each) administered intramuscularly according to the following schedule: A first dose at Month 0 followed by a second dose administered anytime between 2 and 6 months later.
  Interventions: Biological: Shingrix

INTERVENTIONS:
Biological: Shingrix — Biological: SHINGRIX
  SHINGRIX is a vaccine indicated for prevention of herpes zoster (shingles) in adults aged 18 years and older.
  SHINGRIX is a suspension for injection supplied as a single-dose vial of lyophilized glycoprotein e (ge) antigen component to be reconstituted with the accompanying vial of AS01B adjuvant suspension component. A single dose after reconstitution is 0.5 mL.
  Dose and Schedule: Two doses (0.5 mL each) administered intramuscularly according to the following schedule: A first dose at Month 0 followed by a second dose administered anytime between 2 and 6 months later.
  Other Names: Recombinant zoster vaccine

SUMMARY:
Inflammatory bowel disease (IBD) is a chronic inflammatory state of the gastrointestinal tract affecting 1.6-3.1 million people in the United States. Patients with IBD are treated with immunosuppressants that increase their risk of herpes zoster (HZ), also known as shingles.

Those with IBD have a two-fold increased risk for HZ compared to age matched controls. Because most IBD patients are treated with systemic immunosuppressants, which are an independent risk factor for HZ, the live attenuated HZ vaccine was not recommended. However, the release of the new inactivated HZ vaccine, Shingrix (GlaxoSmithKline), presents new opportunities for preventive care.

DETAILED DESCRIPTION:
The purpose of this study is to determine the immunogenicity of the herpes zoster subunit vaccine in inflammatory bowel disease patients on vedolizumab compared to those on anti-tumor necrosis factor (TNF) monotherapy.

The study will evaluate humoral and cell mediated immunity in patients with IBD on vedolizumab who receive the two-dose herpes zoster vaccine. The investigators will evaluate short term, one month after second vaccination dose and sustained immunogenicity at 6 and 12 months post vaccination.

The central hypothesis of this proposal is that IBD patients on vedolizumab should be able to mount a normal vaccine response comparable to those on anti-TNF monotherapy who might benefit from a third dose of the subunit vaccine as has been evaluated in HIV and transplant populations. The hypothesis is that IBD patients on vedolizumab will be able to mount a superior response to those on anti-TNF therapy. A recent study showed that hepatitis B vaccine immunogenicity was not affected by vedolizumab.

The study population will include adult patients aged 18 to 70 with IBD (diagnosed by standard clinical, radiographic, endoscopic, and histopathologic criteria) receiving care at University of Wisconsin Hospital and Clinics. There is no randomization or use of placebo in this study. Two study groups will be established:

* Group A: Patients with IBD on anti-TNF monotherapy
* Group B: Patients with IBD on vedolizumab monotherapy

Eligible patients with IBD will be recruited from the University of Wisconsin Hospital and Clinics.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is between the ages of 18-70 years, inclusive.
2. History of primary varicella infection (chicken pox) Confirmed by a previous history of positive varicella zoster virus (VZV) Immunoglobulin G antibody or history of chicken pox
3. Patient has a history of ulcerative colitis (UC) or Crohn's disease diagnosed by standard clinical, radiographic, endoscopic, and histopathologic criteria.
4. Patient is receiving one of the following treatments for their IBD Group A: Anti-TNF monotherapy (adalimumab, certolizumab, golimumab, infliximab) Group B: Vedolizumab monotherapy
5. Patient has been on stable treatment for IBD for at least three months.

Exclusion Criteria:

1. Previous receipt of any HZ vaccine
2. Allergy to zoster vaccine or a component of it
3. Other underlying chronic medical condition that could affect immunogenicity to vaccines (rheumatoid arthritis, etc.)
4. History of herpes zoster or post herpetic neuralgia within the past year.
5. Patient cannot or will not provide written informed consent.
6. Patient is being administered immunomodulators currently or within the past three months
7. Patient has been taking any dose of oral or intravenous steroids within 30 days prior to immunization.
8. Patient has received polyclonal immunoglobulin therapy or blood products within the last year.
9. Patient is pregnant per self-reporting or older than age 70 years
10. Unable to provide appropriate informed consent due to being illiterate or impairment in decision-making capacity.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2023-10-12 (Actual); Study Completion 2024-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Freddy Caldera, DO, Principal Investigator — UW School of Medicine and Public Health
Locations (1):
- University of Wisconsin Digestive Health Center, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Caldera F, Mogallapalli H, Abusalim AR, Farraye FA, Hayney MS. Immunogenicity and Safety of Recombinant Herpes Zoster Vaccine in Patients With Inflammatory Bowel Disease on Vedolizumab or Anti-Tumor Necrosis Factor Therapy. Clin Transl Gastroenterol. 2025 Nov 1;16(11):e00924. doi: 10.14309/ctg.0000000000000924. PMID 40995992

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at UW Health from May 2019 to July 2023
Groups:
- Vedolizumab: Patients with IBD on vedolizumab monotherapy will be given the shingrix vaccine.
  Dose and Schedule: Two doses (0.5 mL each) administered intramuscularly according to the following schedule: A first dose at Month 0 followed by a second dose administered anytime between 2 and 6 months later.
  Shingrix: Biological: SHINGRIX
  SHINGRIX is a vaccine indicated for prevention of herpes zoster (shingles) in adults aged 18 years and older.
  SHINGRIX is a suspension for injection supplied as a single-dose vial of lyophilized glycoprotein e (ge) antigen component to be reconstituted with the accompanying vial of AS01B adjuvant suspension component. A single dose after reconstitution is 0.5 mL.
- Anti-TNF Monotherapy: Patients with IBD on Anti-TNF monotherapy will be given the shingrix vaccine.
  Dose and Schedule: Two doses (0.5 mL each) administered intramuscularly according to the following schedule: A first dose at Month 0 followed by a second dose administered anytime between 2 and 6 months later.
  Shingrix: Biological: SHINGRIX
  SHINGRIX is a vaccine indicated for prevention of herpes zoster (shingles) in adults aged 18 years and older.
  SHINGRIX is a suspension for injection supplied as a single-dose vial of lyophilized glycoprotein e (ge) antigen component to be reconstituted with the accompanying vial of AS01B adjuvant suspension component. A single dose after reconstitution is 0.5 mL.
Period: Overall Study
Arm/Group | Vedolizumab | Anti-TNF Monotherapy
Started | 16 | 17
Received First Dose | 15 | 17
Received Second Dose | 15 | 15
Completed 90 Day Follow Up | 15 | 15
Completed 1 Year Follow Up | 14 | 15
Analyzed | 15 | 15
Completed | 14 | 15
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vedolizumab | Anti-TNF Monotherapy | Total
Number analyzed (Participants) | 16 | 17 | 33
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 55 [41 to 65] | 62 [54 to 62] | 58 [48 to 62.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 4 | 13
  Male | 7 | 13 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 15 | 17 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 16 | 16 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 17 | 33
Smoking Status [Count of Participants; unit: Participants]
  Former Smoker | 4 | 6 | 10
  Current Smoker | 1 | 1 | 2
Participants with Crohn's Disease [Count of Participants; unit: Participants] | 8 | 14 | 22
Current Irritable Bowel Disease (IBD) Medication [Count of Participants; unit: Participants]
  Adalimumab | 0 | 9 | 9
  Infliximab | 0 | 5 | 5
  Certolizumab | 0 | 3 | 3
  Vedolizumab | 16 | 0 | 16
  Sulfasalazine | 0 | 0 | 0
Previous IBD Medications [Count of Participants; unit: Participants]
  Previous anti-TNF | 13 | 0 | 13
  5-ASA | 12 | 4 | 16
  Methotrexate or azathioprine | 9 | 4 | 13
Positive history of herpes zoster [Count of Participants; unit: Participants] | 2 | 4 | 6
Length of disease [Median (Inter-Quartile Range); unit: months] | 162 [69 to 356] | 344 [141 to 476] | 243 [106 to 409]
Previous IBD surgery [Count of Participants; unit: Participants] | 2 | 12 | 14
Steroid use in past year [Count of Participants; unit: Participants] | 6 | 2 | 8
Charlson Comorbidity Score [Median (Inter-Quartile Range); unit: units on a scale] — None: score 0 Mild: scores of 1-2 Moderate: scores of 3-4 Severe: scores of 5 or higher (up to 37)
  units on a scale | 1.5 [0 to 3.75] | 3 [1 to 4] | 2.1 [0.5 to 3.8]

OUTCOME MEASURES:

1. Primary Outcome: Change in Cell Mediated Immunity
Description: The primary objective will be the change in cell mediated immunity (CMI) as measured by ELISPOT from pre-immunization to one month after receiving second dose of vaccine.
Time Frame: It will be measured from pre-immunization to 1 month after receiving second dose of booster vaccine post-immunization.
Measure: Median (Inter-Quartile Range); unit: cells per million
Arm/Group | Vedolizumab | Anti-TNF Monotherapy
Number analyzed (Participants) | 15 | 15
cells per million
  Pre-Vaccine | 33 [5 to 58] | 33 [13 to 88]
  One month after series completion of two dose series | 33 [17 to 91] | 50 [36 to 193]
Statistical Analysis 1: Comparison: Vedolizumab vs Anti-TNF Monotherapy; one month after series completion of two dose series; Test type: Superiority; p = 0.16, Mann-Whitney U test

2. Secondary Outcome: Percent of Participants With Sustained Cell Mediated Immunity Measured Via ELISPOT After Immunization.
Description: Sustained change in CMI at 6 months will be assessed after receiving a second dose of booster vaccine post-immunization. CMI will be measured via ELISPOT
Time Frame: Baseline to 6 months post-immunization 2nd dose of vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Vedolizumab | Anti-TNF Monotherapy
Number analyzed (Participants) | 15 | 15
Participants | 15 | 15

3. Secondary Outcome: Percent of Participants With a Change in Antibody Concentration Post Immunization
Description: A secondary outcome will be the change in varicella zoster virus (VZV) antibody concentration comparing pre-immunization to post immunization antibody concentration.
Time Frame: pre-immunization to one month 2nd dose post-immunization
Measure: Count of Participants; unit: Participants
Arm/Group | Vedolizumab | Anti-TNF Monotherapy
Number analyzed (Participants) | 15 | 15
Participants | 15 | 15

4. Secondary Outcome: Percent of Participants With a Change in Antibody Concentration That is Sustained at 6 Months
Description: Sustained change in VZV antibody concentration at 6 months after receiving a second dose of booster vaccine post-immunization will be assessed.
Time Frame: Baseline to 6 months post-immunization
Measure: Count of Participants; unit: Participants
Arm/Group | Vedolizumab | Anti-TNF Monotherapy
Number analyzed (Participants) | 15 | 15
Participants | 15 | 15

5. Secondary Outcome: Number of Participants Who Experienced Vaccine Related Adverse Events After Dose 1
Description: To evaluate for adverse effects following immunization patients will receive phone calls from study personnel to ascertain vaccine-related adverse effects.
  Dose and Schedule: Two doses (0.5 mL each) administered intramuscularly according to the following schedule: A first dose at Month 0 followed by a second dose administered anytime between 2 and 6 months later.
Time Frame: Dose 1 (Month 0)
Measure: Count of Participants; unit: Participants
Groups:
- Vedolizumab Dose 1: Grade 1: Grade 1 (Mild) Adverse Event
  Patients with IBD on vedolizumab monotherapy will be given the shingrix vaccine.
- Vedolizumab Dose 1: Grade 2: Grade 2 (Moderate) Adverse Event
  Patients with IBD on vedolizumab monotherapy will be given the shingrix vaccine.
- Vedolizumab Dose 1: Grade 3: Grade 3 (Severe) Adverse Event
  Patients with IBD on vedolizumab monotherapy will be given the shingrix vaccine.
- Vedolizumab Dose 1: Grade 4: Grade 4 (Life Threatening) Adverse Event
  Patients with IBD on vedolizumab monotherapy will be given the shingrix vaccine.
- Anti-TNF Monotherapy Dose 1: Grade 1: Grade 1 (Mild) Adverse Event
  Patients with IBD on Anti-TNF monotherapy will be given the shingrix vaccine.
- Anti-TNF Monotherapy Dose 1: Grade 2: Grade 2 (Moderate) Adverse Event
  Patients with IBD on Anti-TNF monotherapy will be given the shingrix vaccine.
- Anti-TNF Monotherapy Dose 1: Grade 3: Grade 3 (Severe) Adverse Event
  Patients with IBD on Anti-TNF monotherapy will be given the shingrix vaccine.
- Anti-TNF Monotherapy Dose 1: Grade 4: Grade 4 (Life Threatening) Adverse Event
  Patients with IBD on Anti-TNF monotherapy will be given the shingrix vaccine.
Arm/Group | Vedolizumab Dose 1: Grade 1 | Vedolizumab Dose 1: Grade 2 | Vedolizumab Dose 1: Grade 3 | Vedolizumab Dose 1: Grade 4 | Anti-TNF Monotherapy Dose 1: Grade 1 | Anti-TNF Monotherapy Dose 1: Grade 2 | Anti-TNF Monotherapy Dose 1: Grade 3 | Anti-TNF Monotherapy Dose 1: Grade 4
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 15 | 15 | 15
Participants
  Any Systemic Adverse Effect | 7 | 1 | 0 | 0 | 6 | 0 | 0 | 0
  Headaches | 6 | 0 | 0 | 0 | 3 | 0 | 0 | 0
  Plugged ear | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Intermittent fever/chills | 3 | 0 | 0 | 0 | 2 | 0 | 0 | 0
  Lymphadenopathy | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Congestion | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Fatigue | 5 | 0 | 0 | 0 | 2 | 0 | 0 | 0
  Myalgias/joint pain | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0
  Any Local Adverse Effect | 8 | 1 | 0 | 0 | 11 | 2 | 0 | 0
  Pain/Soreness | 9 | 1 | 0 | 0 | 12 | 1 | 0 | 0
  Pruritus | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Erythema | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0
  Swelling | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Warmth | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants Who Experienced Vaccine Related Adverse Events After Dose 2
Description: as for outcome 5
Time Frame: Dose 2 (anytime from Month 2 to Month 6)
Measure: Count of Participants; unit: Participants
Groups:
- Vedolizumab Dose 2: Grade 1: Grade 1 (Mild) Adverse Event
  Patients with IBD on vedolizumab monotherapy will be given the shingrix vaccine.
- Vedolizumab Dose 2: Grade 2: Grade 2 (Moderate) Adverse Event
  Patients with IBD on vedolizumab monotherapy will be given the shingrix vaccine.
- Vedolizumab Dose 2: Grade 3: Grade 3 (Severe) Adverse Event
  Patients with IBD on vedolizumab monotherapy will be given the shingrix vaccine.
- Vedolizumab Dose 2: Grade 4: Grade 4 (Life Threatening) Adverse Event
  Patients with IBD on vedolizumab monotherapy will be given the shingrix vaccine.
- Anti-TNF Monotherapy Dose 2: Grade 1: Grade 1 (Mild) Adverse Event
  Patients with IBD on Anti-TNF monotherapy will be given the shingrix vaccine.
- Anti-TNF Monotherapy Dose 2: Grade 2: Grade 2 (Moderate) Adverse Event
  Patients with IBD on Anti-TNF monotherapy will be given the shingrix vaccine.
- Anti-TNF Monotherapy Dose 2: Grade 3: Grade 3 (Severe) Adverse Event
  Patients with IBD on Anti-TNF monotherapy will be given the shingrix vaccine.
- Anti-TNF Monotherapy Dose 2: Grade 4: Grade 4 (Life Threatening) Adverse Event
  Patients with IBD on Anti-TNF monotherapy will be given the shingrix vaccine.
Arm/Group | Vedolizumab Dose 2: Grade 1 | Vedolizumab Dose 2: Grade 2 | Vedolizumab Dose 2: Grade 3 | Vedolizumab Dose 2: Grade 4 | Anti-TNF Monotherapy Dose 2: Grade 1 | Anti-TNF Monotherapy Dose 2: Grade 2 | Anti-TNF Monotherapy Dose 2: Grade 3 | Anti-TNF Monotherapy Dose 2: Grade 4
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15 | 15 | 15 | 15
Participants
  Any Systemic Adverse Effect | 5 | 1 | 2 | 0 | 3 | 3 | 0 | 0
  Headaches | 3 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  Plugged ear | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Intermittent fever/chills | 4 | 0 | 1 | 0 | 1 | 2 | 0 | 0
  Lymphadenopathy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Congestion | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Fatigue | 4 | 1 | 0 | 0 | 1 | 1 | 0 | 0
  Myalgias/joint pain | 6 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  Any Local Adverse Effect | 10 | 0 | 0 | 0 | 7 | 1 | 0 | 0
  Pain/Soreness | 8 | 0 | 0 | 0 | 6 | 1 | 0 | 0
  Pruritus | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Erythema | 4 | 0 | 0 | 0 | 2 | 0 | 0 | 0
  Swelling | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Warmth | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants Experiencing a Change in Disease Activity Post Immunization Reported
Description: The Simple Clinical Colitis Activity Index (SCCAI) will be used to measure disease activity. It is a questionnaire with six subscore topics with scores defined by UC signs and symptoms from 0 to 4 for a range of scores from 0 to 17. Total scores are interpreted as: Remission = score of 0 to 4 points, Mild Activity = score of 5 to 7 points, Moderate Activity = Score of 8 to 16 points, and Severe Activity = Score of > 16 points. Number of participants experiencing a change will be reported.
Time Frame: at the baseline visit and one month after receipt of each vaccine
Measure: Count of Participants; unit: Participants
Arm/Group | Vedolizumab | Anti-TNF Monotherapy
Number analyzed (Participants) | 15 | 15
Participants
  baseline | 0 | 0
  1 month post-dose 1 | 0 | 0
  1 month post-dose 2 | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 12 months post second dose (approximately 425 days on study)
Description: data collected via phone call and follow up visits (follow up phone call at day 12, visit at day 60, phone call at day 72, visit at day 90 (one month post-second-dose), visit at day 240 (6 months post-second-dose), visit at day 425 (12 months post-second-dose)
Groups:
- Vedolizumab: Dose 1; Vedolizumab: Dose 2: Patients with IBD on vedolizumab monotherapy will be given the shingrix vaccine.
  Dose and Schedule: Two doses (0.5 mL each) administered intramuscularly according to the following schedule: A first dose at Month 0 followed by a second dose administered anytime between 2 and 6 months later.
- Anti-TNF Monotherapy: Dose 1; Anti-TNF Monotherapy: Dose 2: Patients with IBD on Anti-TNF monotherapy will be given the shingrix vaccine. Dose and Schedule: Two doses (0.5 mL each) administered intramuscularly according to the following schedule: A first dose at Month 0 followed by a second dose administered anytime between 2 and 6 months later.
- Vedolizumab: 6 Months Post Follow up; Vedolizumab: 12 Months Post Follow up: Patients with IBD on vedolizumab monotherapy will be given the shingrix vaccine.
- Anti-TNF Monotherapy: 6 Months Post Follow up; Anti-TNF Monotherapy: 12 Months Post Follow up: Patients with IBD on Anti-TNF monotherapy will be given the shingrix vaccine.
Arm/Group | Vedolizumab: Dose 1 | Anti-TNF Monotherapy: Dose 1 | Vedolizumab: Dose 2 | Anti-TNF Monotherapy: Dose 2 | Vedolizumab: 6 Months Post Follow up | Anti-TNF Monotherapy: 6 Months Post Follow up | Vedolizumab: 12 Months Post Follow up | Anti-TNF Monotherapy: 12 Months Post Follow up
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15 | 0/15 | 0/15 | 0/14 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15 | 0/15 | 0/15 | 0/14 | 0/15
Other Adverse Events (participants affected / at risk) | 10/15 | 13/15 | 10/15 | 7/15 | 0/15 | 0/15 | 0/14 | 0/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vedolizumab: Dose 1 (N=15) | Anti-TNF Monotherapy: Dose 1 (N=15) | Vedolizumab: Dose 2 (N=15) | Anti-TNF Monotherapy: Dose 2 (N=15) | Vedolizumab: 6 Months Post Follow up (N=15) | Anti-TNF Monotherapy: 6 Months Post Follow up (N=15) | Vedolizumab: 12 Months Post Follow up (N=14) | Anti-TNF Monotherapy: 12 Months Post Follow up (N=15)
Headache (General disorders) | 6 | 3 | 3 | 2 | 0 | 0 | 0 | 0
Plugged Ear (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intermittent Fever or Chills (General disorders) | 3 | 2 | 5 | 3 | 0 | 0 | 0 | 0
Lymphadenopathy (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Congestion (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 5 | 2 | 5 | 2 | 0 | 0 | 0 | 0
Myalgias or Joint Pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 7 | 1 | 0 | 0 | 0 | 0
Pain or Soreness (Skin and subcutaneous tissue disorders) | 10 | 13 | 8 | 7 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 3 | 4 | 2 | 0 | 0 | 0 | 0
Swelling (Skin and subcutaneous tissue disorders) | 3 | 1 | 2 | 1 | 0 | 0 | 0 | 0
Warmth (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-16): https://cdn.clinicaltrials.gov/large-docs/91/NCT03798691/Prot_SAP_000.pdf